CLINICAL TRIAL: NCT07329205
Title: Effects of Femoral Nerve Mobilization on Pain Intensity, Function, Quality of Life and Central Sensitization in Patients With Knee Osteoarthritis
Brief Title: Femoral Nerve Mobilization for Patients With Knee Osteoarthritis
Acronym: RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Mohammad Moustafa Aldosoukki Hegazy, assisstant professor , department of health and rehabilitation sciences, college of applied medical siences, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/025/015
Record Dates: First submitted 2025-12-15; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthristis
Keywords: NEURAL MOBILIZATION; Knee osteoarthritis; conventional physical therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Traditional physical therapy
  Interventions: Other: traditional physical therapy
- Neural mobilization group (Experimental): traditional physical therapy plus femoral nerve mobilization
  Interventions: Other: traditional physical therapy; Other: Femoral nerve mobilization

INTERVENTIONS:
Other: traditional physical therapy — stretching exercises for hamstring, calf muscles and iliotibial band in addition to isotonic exercise for hip extensors and abductors and isometric quadriceps exercise
Other: Femoral nerve mobilization — A physiotherapist guided the patients in performing active mobilization of the femoral nerve. The prescribed method for active neural mobilization involved assuming a prone position supported by the forearms with a slight extension of the spine, flexion of the knee, and extension of the cervical spine. This was followed by performing the opposite movement
  Arms: Neural mobilization group

SUMMARY:
Background: Knee osteoarthritis (KO) is considered as a cause of disability among the elderly, causing pain, reduced quality of life, and decreased functionality. There is a limited knowledge about using femoral nerve mobilization in treating patients with arthritic changes.

Objectives: This study will be designed to determine the efficacy of adding of femoral nerve mobilization on pain intensity, function, quality of life and central sensitization in patients with knee osteoarthritis Methods: Thirty patients (aged ≥50 years with KO Kellgren-Lawrence grades I-II) will be included in this study: Patients will randomly be assigned into two groups: group A will receive traditional physical therapy while group B will receive femoral nerve mobilization in addition to traditional physical therapy. Three sessions will be performed for four weeks by 3 session /week. Patients will be evaluated for pain intensity using the numerical rating scale (NRS), knee function by WOMAC scale, quality of life by 12-item Short Form Survey questionnaire (SF-12) and central sensitization by the Arabic version of central sensitization inventory (CSI).

ELIGIBILITY:
Inclusion Criteria:

* patients aged 50 years or older, diagnosed with KO according to theAmerican College of Rheumatology's criteria with knee pain, and grade I or II on the Kellgren-Lawrence radiographic scale

Exclusion Criteria:

* individuals suffering from chronic conditions considered to be perpetuating factors (e.g., fibromyalgia)
* those with conditions causing lower extremity pain
* individuals who had taken analgesics within 24 h before evaluations
* those who had undergone corticosteroid or local anesthetic infiltration in the year prior to the study or during the follow-up period
* those using substances that could interfere with treatment
* those with a previous diagnosis of neuropathy (lumbosacral plexus) or myopathy
* those with contraindications to mobilization or exercise, and those with cognitive deficits (dementia, Alzheimer's).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
pain intensity | after 4 weeks
  The pain was assessed by the numerical rating scale (NRS) where zero indicating no pain and 10 indicating maximal pain
central sensitization | after 4 weeks
  The CSI is a validated questionnaire designed to identify symptoms associated with central sensitization. It has two components: Scale A assesses 25 common symptoms in individuals with central sensitization, resulting in a score ranging from 0 to 100. This score was interpreted as follows: subclinical (0-29), mild (30-39), moderate (40-49), severe (50-59), and extreme (60-100). Scale B, which is not scored, collects information on previous diagnoses of specific diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Sattam bin Abdulaziz University, Al Kharj, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pedersini P, Valdes K, Cantero-Tellez R, Cleland JA, Bishop MD, Villafane JH. Effects of Neurodynamic Mobilizations on Pain Hypersensitivity in Patients With Hand Osteoarthritis Compared to Robotic Assisted Mobilization: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2021 Feb;73(2):232-239. doi: 10.1002/acr.24103. Epub 2021 Jan 3. PMID 31675184
- [Result] Yamasaki T, Nakajima H. [Glycogenosis type VII (glycogen storage disease type VII, human muscle-phosphofructokinase deficiency, Tarui's disease)]. Ryoikibetsu Shokogun Shirizu. 2001;(36):28-34. No abstract available. Japanese. PMID 11596390
- [Result] Franklin-Tong VE. Signaling in pollination. Curr Opin Plant Biol. 1999 Dec;2(6):490-5. doi: 10.1016/s1369-5266(99)00017-5. PMID 10607651